CLINICAL TRIAL: NCT04105686
Title: Growth and Tolerance of Young Infants Fed Milk-Based Infant Formula With Oligosaccharides
Brief Title: Growth and Tolerance of Young Infants Fed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL31A
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Growth and Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Infant Formula (Active Comparator): Milk-based study product
  Interventions: Other: Control Infant Formula
- Experimental Infant Formula (Experimental): Milk-based study product with oligosaccharides
  Interventions: Other: Experimental Infant Formula
- Reference Group (No Intervention): Human milk-fed group

INTERVENTIONS:
Other: Control Infant Formula — Ready to feed infant formula, feed ad libitum
  Arms: Control Infant Formula
Other: Experimental Infant Formula — Ready to feed infant formula, feed ad libitum
  Arms: Experimental Infant Formula

SUMMARY:
This is a randomized, multicenter, controlled, double-blind, parallel study to evaluate growth and tolerance of healthy term infants fed milk-based infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health as determined from participant's medical history.
* Participant is a singleton from a full-term birth with a gestational age of 37-42 weeks.
* Participant's birth weight was > 2490 g (~5 lbs. 8 oz.).
* Parent(s) who elect to formula-feed the participant, confirm their intention to feed their infant the study product as the sole source of feeding during the study.
* Parent(s) who elect to feed the participant human milk, confirm their intention to exclusively feed human milk as the sole source of feeding during the study.
* Parent(s) of formula-fed infants confirm their intention not to administer vitamin or mineral supplements, (except for vitamin D supplements), solid foods or juices to their infant from enrollment through the duration of the study.
* Parent(s) of human milk-fed infants confirm their intention not to administer solid foods or juices to their infant from enrollment through the duration of the study (vitamins and minerals are acceptable).
* Participant's parent(s) has voluntarily signed and dated an ICF, approved by an IRB/IEC and provided HIPAA (or applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Participant is taking and plans to continue taking medications (including over the counter), prebiotics, probiotics, home remedies, herbal preparations or rehydration fluids that might affect GI tolerance.
* Participant participates in another study that has not been approved as a concomitant study.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 366 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Weight | Day of life 14 to Day of life 119
  Weight gain per day

SECONDARY OUTCOMES:
Stool Characteristics | Study Day 1 to Day of life 119
  Parent completed diary
Formula Tolerance | Study Day 1 to Day of life 119
  Parent completed diary
Length | Day of life 14 to Day of life 119
  Length gain per day
Head Circumference (HC) | Day of life 14 to Day of life 119
  HC gain per day

OTHER OUTCOMES:
Infant and Household Characteristics | Study Day 1 to Day of Life 119
  Parent reported lifestyle and illness questions
Infant Feeding and Stool Patterns Questionnaire | Exit or Day of life 119
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled in the negative direction
Infant Behavior Questionnaire | Exit or Day of life 42 to Day of life 119
  Parent completed questionnaire; 22 questions with 5-point Likert scale questions, scaled in the negative direction
Formula Satisfaction Questionnaire | Exit or Day of life 119
  Parent completed questionnaire; 12 questions with 5-point Likert scale questions scaled in the negative direction

CONTACTS AND LOCATIONS:
Overall Officials: Timberly Williams, PhD, Study Chair — Abbott Nutrition
Locations (32):
- United States (32):
  - Central Research Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Visions Clinical Research, Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - TOPAZ Clinical Research, Inc., Apopka, Florida
  - University Clinical Research-Deland, LLC dba Avail Clinical Research- West Volusia Pediatrics, DeLand, Florida
  - Children's Research, LLC, Lake Mary, Florida
  - New Horizon Research Center, Miami, Florida
  - Pediatric & Adult Research Center, Orlando, Florida
  - Asclepes Research Centers, Spring Hill, Florida
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - PAS Research, LLC, Tampa, Florida
  - Tekton Research, Chamblee, Georgia
  - Saltzer Health, Nampa, Idaho
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Springs Medical Research, Owensboro, Kentucky
  - Meridian Clinical Research 3080, Baton Rouge, Louisiana
  - Meridan Clinical Research, Omaha, Nebraska
  - Wake Research - Clinical Research Center of Nevada, Las Vegas, Nevada
  - ClinOhio Research Services, Columbus, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Institute of Clinical Research, LLC, Mentor, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Midsouth Center for Clinical Research, Memphis, Tennessee
  - Medical Research Center of Memphis, Memphis, Tennessee
  - Gadolin Research, LLC, Beaumont, Texas
  - Women's Hospital at Renaissance - Doctors Hospital at Renaissance, Edinburg, Texas
  - Mercury Clincial Research, Inc., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Aspen Clinical Research LLC, Orem, Utah
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No